CLINICAL TRIAL: NCT04498429
Title: Effect of Integrated Manual and Verbal Cueing on Functional Transfers in Chronic Stroke Survivors: A Randomized Controlled Study
Brief Title: Effect of Integrated Cueing on Functional Transfers in Chronic Stroke Survivors
Acronym: EOIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Eric Johnson, Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5200090
Record Dates: First submitted 2020-07-28; First posted 2020-08-04 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Hemiplegia and/or Hemiparesis Following Stroke
Keywords: Facilitation; Sit-to-Stand; Manual Cueing; Verbal Cueing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Manual and Verbal Cueing Group (Experimental): A series of 40 training repetitions of sit to stand using the Integrated/Manual Cueing intervention.
  Interventions: Other: Integrated Cueing Protocol
- Verbal Cueing Group (Experimental): A series of 40 training repetitions of sit to stand using the Verbal Cueing intervention
  Interventions: Other: Verbal Cueing Protocol

INTERVENTIONS:
Other: Integrated Cueing Protocol — The first 5 repetitions will include part to whole task practice of partial sit to stand using scripted verbal cueing to facilitate understanding of the task. The goal is to improve midline orientation and alignment during the task of moving from sitting to standing. In addition to verbal cueing, the manual cueing group will receive hands-on tactile facilitation from a trained physical therapist to facilitate appropriate midline weight shift during the sit to stand activity for the series of 40 training repetitions.
  Other Names: Manual Cueing Protocol
  Arms: Integrated Manual and Verbal Cueing Group
Other: Verbal Cueing Protocol — The first 5 repetitions will include part to whole task practice of partial sit to stand using scripted verbal cueing to facilitate understanding of the task. The goal is to improve midline orientation and alignment during the task of moving from sitting to standing. The verbal cueing protocol consists of verbal cueing from a trained physical therapist to facilitate appropriate midline weight shift during the sit to stand activity for the series of 40 training repetitions.
  Arms: Verbal Cueing Group

SUMMARY:
Physical therapists frequently use manual cueing as a tool to improve movement quality in persons recovering from stroke but evidence to support its effectiveness is lacking.

The purpose of this graduate student research study is to determine the immediate and carryover effects of an integrated verbal and manual facilitation approach used by physical therapists during sit to stand training on the midline alignment, muscle activation and quality of movement in chronic stroke survivors with hemiplegia.

DETAILED DESCRIPTION:
Over the last few decades, the profession of physical therapy has heavily relied on manual facilitation to improve motor control and functional movement in persons recovering from stroke or other neurological impairments. In the 1950's, Berta Bobath created Neuro-Developmental Treatment (NDT), a systematic problem-solving approach that is one of the most widely used methodologies in neurorehabilitation. NDT relies heavily on verbal and tactile facilitation as an integrated approach to improve motor control in persons with hemiplegia. However, current systematic reviews have stated that adequate evidence for the effectiveness of neuro facilitation is lacking. In the current climate of evidence-based practice, neurologic physical therapists no longer blindly accept the use of traditional interventions and instead rely on peer-reviewed research studies to support their clinical decision-making.

However, the question remains for many physical therapists: are skilled manual cues really an essential ingredient in the post-stroke recipe? Most practicing neurologic physical therapists would claim that their hands are their most valuable tools and that the way in which they use their hands has a direct effect on movement patterns and functional outcomes with their patients. Ploughman and colleagues reported that manual tactile cues during gait had "robust but short-lived impacts on cadence and time in double support" during gait but their findings are merely a step in the right direction. An integrative approach of both manual and verbal cues have anecdotally shown to be effective to treat impairments from stroke but there continues to be a dearth of evidence to accurately support the pervasive use of manual facilitation by physical therapists. While support for manual tactile cueing is merely beginning to move in the right direction, strong evidence exists that task specific training can improve functional outcomes by focusing training on desired movements and activities. But what part does manual cueing truly play in task specific training? Sit to stand is an essential activity of daily living that is often impaired in stroke survivors and is commonly trained by physical therapists from both task specific training and NDT schools of thought. Physical therapists need further clarification as to which methods are most effective for facilitating maximum learning and recovery during this functional task in order to craft an ideal recipe.

Training correct movement patterns in order to improve functional independence is important at every stage of recovery after stroke. Kerr et al. suggested that successful sit to stand movements require proper training of the critical timing of events as well as improving synergistic activation of the appropriate lower limb musculature. Ultimately, asymmetry can lead to a conditioned suppression of available movement termed "learned non-use". Continual reinforcement of poor movement strategies thus leads to passive suppression of maximally efficient normal movements unless the stroke survivor is actively retrained to unlock masked abilities over time. Teasell and colleagues confirmed the importance of skilled rehabilitation throughout all phases of recovery including the chronic stroke phase, though this important population regularly experiences fewer opportunities to participate in therapy as time progresses. Measurable gains may be slower at this stage but the ability to perform essential mobility tasks remains just as important to the individual.

Thus, the purpose of this graduate student research study is to determine the immediate and carryover effects of an integrated verbal and manual facilitation approach during sit to stand training on the midline alignment, muscle activation and quality of movement in chronic stroke survivors with hemiplegia. By determining the essential ingredients that lead to an ideal recipe for success, physical therapists may have more evidence-based tools available to maximize the independence, quality of life and confidence of their patients.

Procedures: Session 1: All participants will complete the initial paperwork and then be randomized into Verbal Cueing Group or Verbal + Manual Cueing Group using envelopes that are predetermined from a random number table. Height will be assessed using a stadiometer and weight using a scale. Subjects will then have trajectory markers and surface electromyographic (EMG) sensors placed according to the chart. This includes 24 individual marker trajectories, two thigh clusters and two shank clusters of four trajectories each for a total of 40 markers and 6 surface EMG sensors that will be placed on major muscle groups of the lower extremities. Once the setup has been completed and verified, the subject will perform two static standing trials, followed by two initial sit to stand (STS) trials to determine their baseline variables. This format will be followed by both the Verbal Cueing and the Verbal + Manual Cueing throughout the treatment session. The first 5 repetitions of both groups will include part to whole task practice of partial sit to stand using scripted verbal cueing to facilitate understanding of the task. The goal of both groups is to improve midline orientation and alignment during the task of moving from sitting to standing.

After the first 5 repetitions, the subject will perform two sit to stand trials on their own following the clinician's scripted verbal commands. Next, five Manual + Verbal Cueing or Verbal Cueing trials will commence followed by another two PostCue trials. This repeated sequence of 5 cued trials followed by 2 assessment trials will continue for a total of 40 sit to stand trials. After a 5-minute rest period the subject will then be asked to perform two additional STS to determine retention of learning over that interval. Next, two isometrically resisted sit to stand trials will be performed for EMG normalization. Once the EMG normalization is completed, the subject will then be told they are done and may get up to leave. When they get up to leave, their sit to stand activity will also be discretely recorded for comparison to their last knowingly observed trial. This is based on the Actual Amount of Use Test (AAOUT) in which subjects are observed under normal circumstances to assess whether the learning was integrated into functional use when the subject doesn't think they are being observed.

At the end of session #1, the investigator will ask the subject what strategy most helped them achieve midline. Based on their feedback, the investigator will create and issue a home exercise program (HEP) handout that incorporates that subjective report. Examples include statements such as, "Feeling the pressure through my left leg" or "Leaning to my left". This cue will be placed on a brightly colored card that will be placed near where the subject practices sitting to standing most often in their home environment. The card will also contain an easy to mark log to encourage practice of the STS task over the next 3-5 days. The subject will be instructed to perform the exercises at the times specified on the card using the subject's subjective to help encourage maximal midline orientation. Permission will be obtained to text the subject on a regular basis to remind them to perform the exercises.

Session 2: Participants who choose to return will come back within 3 to 5 days of Session #1. Subjects will be asked to bring their HEP card to verify compliance via the practice log. After placement of the trajectory markers (but not the EMG), subjects will be asked to perform two trials of sit to stand, regardless of their original group. They will then be assessed with the AAOUT test in the same manner as the end of session #1. Afterward, participants in the Verbal Cueing group will be offered the Integrated Cueing approach if they so choose.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Right CVA with left hemiplegia > 6 Months
* Able to ambulate with no more than help than supervision
* Must be able to stand without an assistive device or ankle foot orthosis
* Must be able to follow two-step verbal commands

Exclusion Criteria:

* History of injury from a recent fall within the last 3 months
* Currently participating in rehabilitation during the time frame of their participation in this study
* Additional musculoskeletal or neurological conditions that may impair ability to perform sit to stand safely

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
Midline Orientation via Symmetry Ratio | Baseline and immediately after the intervention
  The participant's ability to equally distribute their weight throughout the sit to stand task will be measured via two force plates integrated with the Qualisys motion capture system. The ratio is calculated via dividing the weight on the hemiparetic leg by the weight on the non-hemiparetic side. A score of 1 indicates equal weight bearing.
Midline Orientation via Trunk Lateral Lean angle | Baseline and immediately after the intervention
  The participant's ability to maintain an upright trunk throughout the sit to stand task as measured by computations from the Qualisys motion capture system using 40 trajectory markers. Perfect midline orientation would be a value of 0 degrees indicating midline orientation.
Muscle Activation | During after the intervention
  Comparison of muscle activation between normal and hemiparetic lower extremity extensor muscle groups as measured with surface electromyography (EMG) and processed through the Qualisys motion capture system. Change will be indicated by subtracting max contraction per various extensor muscle groups as a composite measure during the activity from initial max contraction of the same muscle group.
Time to complete Sit to Stand Activity | Baseline and immediately after the intervention
  A measurement of the total elapsed time to perform the sit to stand activity as measured from initial movement to highest position of center of mass

CONTACTS AND LOCATIONS:
Overall Officials: Eric G Johnson, DSc, Principal Investigator — Loma Linda University
Locations (2):
- United States (2):
  - Loma Linda University Health, Loma Linda, California
  - Loma Linda University, Loma Linda, California

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared